CLINICAL TRIAL: NCT01316445
Title: Comparing the Pharmacodynamics of Nasal and Buccal Midazolam Using EEG
Brief Title: Pharmacodynamics of Nasal and Buccal Midazolam Using EEG
Acronym: nMDZ-EEG
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Funding agency no longer provide support.
Sponsor: Columbia University (Other)
Collaborators: Upsher-Smith Laboratories (Industry)
Responsible Party: Principal Investigator, Bin Tu, Associate Research Scientist, Columbia University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AAAF3704
Record Dates: First submitted 2011-03-15; First posted 2011-03-16 (Estimated); Last update posted 2015-02-04 (Estimated); Status verified 2015-02

CONDITIONS: Epilepsy
Keywords: Electroencephalography; Benzodiazepines; Midazolam
MeSH Terms: conditions — Epilepsy | interventions — Midazolam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- nasal Midazolam (Experimental): 3 mg of the standard IV solution of midazolam (5 mg/mL) was given via a metered-dose nasal sprayer (6 sprays × 0.1 ml/spray, or 6 × 0.5 mg/spray) divided between the two nostrils within 1-2 min. During the EEG, vital signs (blood oxygen saturation, blood pressure, pulse and respiratory rate) were monitored and a nurse and a physician were available at all times. Subjects were monitored for 2 hours after administration of midazolam to ensure adequate recovery from sedation.
  Interventions: Drug: nasal Midazolam

INTERVENTIONS:
Drug: nasal Midazolam — Intranasal and buccal administration of the standard IV formulation of midazolam (5mg/mL), administered via a metered dose sprayer at 0.1mL/spray (i.e. 0.5mg/spray). Administration will be via three sprays in each nostril (for nasal) or three sprays between the cheek and the gum per side (for buccal).
  Other Names: Versed

SUMMARY:
Approximately 3 million individuals suffer from epilepsy in America alone and about 200,000 new cases of epilepsy in America are diagnosed each year (Epilepsy Foundation, 2005). Epilepsy can be defined as a condition in which a person has recurrent, unprovoked seizures. Prolonged or back-to-back repetitive seizures, known as "acute repetitive seizures" (ARS), are medical emergencies. ARS can occur unexpectedly, a circumstance for which quick and efficient antiepileptic drugs are needed for household and prehospital use. Currently, benzodiazepines are the antiepileptic drug of choice when dealing with ARS because they are proven to be efficient and take little time to work. Benzodiazepines can be administered by mouth, by vein via a needle (intravenously; IV), rectally, between the cheek and gum (buccally), or in the nose (intranasally; IN). The nasal formulation is not yet FDA-approved. The rectal treatment route has been commonly used for acute seizure treatment in past years, but recent studies propose that the nasal route for benzodiazepines may be better overall for home treatment and easier to administer (see Wermeling, 2009). For many "out of hospital" situations, nasal benzodiazepines can be more convenient and more comfortable than rectal treatment. In addition to the above benefits, nasal benzodiazepines are rapidly absorbed by the blood vessels in the nose and the time of drug administration and cessation of seizures may thus be reduced using nasal routes. This study sets out to characterize how fast buccal and nasal treatments begin to work on the brain by monitoring brain waves during administration of the drug, and to determine whether nasal or buccal administration is best.

DETAILED DESCRIPTION:
Past out-of-hospital treatments for acute epileptic seizures have met with limited effectiveness, convenience, speed, and safety. The only FDA-approved treatment for acute repetitive seizures must be given rectally, but nasal or buccal midazolam have been shown to be at least as effective. The purpose of this study is to characterize the time to effect on brain activity of intranasal (or nasal) midazolam and compare it with buccal midazolam. This research will recruit patients with epilepsy who are undergoing EEG recordings for clinical purposes, including those with intracranial EEG. EEG will be evaluated during administration of buccal or nasal midazolam for augmentation of beta waves signifying action of midazolam on the brain, and the time to effect will be compared between buccal and nasal formulations. Subjects will be given a brief survey after the administration to evaluate sedation, discomfort and other adverse effects of the medication. This study will help characterize the action of nasal and buccal benzodiazepines and to determine the most effective method of administration.

ELIGIBILITY:
Inclusion Criteria:

* adults undergoing extracranial EEG in an Epilepsy Monitoring Unit
* adults undergoing intracranial EEG in an Epilepsy Monitoring Unit
* adults with chronically implanted intracranial neurostimulators with the capacity for continuous intracranial EEG monitoring

Exclusion Criteria:

* any patient on additional sedative medications (narcotics, other central nervous system depressants)
* any patient with documented sensitivity or adverse reaction to any benzodiazepine

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2011-07; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
25% increase in total beta power for at least 1 minute at 10-30Hz | for 30 mins after administration of drug
  Quantitative and qualitative visual EEG analysis for benzodiazepine-induced beta activity, total power of ~10-30 Hz activity

SECONDARY OUTCOMES:
beta activity at 10-12 Hz | for 30 minutes after drug administration
  Qualitative visual and quantitative EEG analysis for benzodiazepine-induced beta activity at bands of 10-12 Hz
beta activity at 30-40Hz | for 30 minutes after drug administration
  Qualitative visual and quantitative EEG analysis for benzodiazepine-induced beta activity at bands of 30-40Hz.
sedation | for 30 minues after drug administration
  Subject perception of sedation will be evaluated using yes or no type questions, evaluation questions using a visual analogue scale (from 1 to 10) and open response questions.
pain/discomfort | for 30 minutes after drug administration
  Subject perception of discomfort will be evaluated using yes or no type questions, evaluation questions on a visual analogue scale (from 1 to 10), and open-response questions.

CONTACTS AND LOCATIONS:
Overall Officials: Derek Chong, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, Milstein Hospital, New York, New York, United States

REFERENCES:
- [Background] Loftsson T, Gudmundsdottir H, Sigurjonsdottir JF, Sigurdsson HH, Sigfusson SD, Masson M, Stefansson E. Cyclodextrin solubilization of benzodiazepines: formulation of midazolam nasal spray. Int J Pharm. 2001 Jan 5;212(1):29-40. doi: 10.1016/s0378-5173(00)00580-9. PMID 11165818
- [Background] Knoester PD, Jonker DM, Van Der Hoeven RT, Vermeij TA, Edelbroek PM, Brekelmans GJ, de Haan GJ. Pharmacokinetics and pharmacodynamics of midazolam administered as a concentrated intranasal spray. A study in healthy volunteers. Br J Clin Pharmacol. 2002 May;53(5):501-7. doi: 10.1046/j.1365-2125.2002.01588.x. PMID 11994056
- [Background] Wermeling DP, Record KA, Kelly TH, Archer SM, Clinch T, Rudy AC. Pharmacokinetics and pharmacodynamics of a new intranasal midazolam formulation in healthy volunteers. Anesth Analg. 2006 Aug;103(2):344-9, table of contents. doi: 10.1213/01.ane.0000226150.90317.16. PMID 16861415
- [Background] Wermeling DP, Record KA, Archer SM, Rudy AC. A pharmacokinetic and pharmacodynamic study, in healthy volunteers, of a rapidly absorbed intranasal midazolam formulation. Epilepsy Res. 2009 Feb;83(2-3):124-32. doi: 10.1016/j.eplepsyres.2008.10.005. Epub 2008 Nov 29. PMID 19046855
- [Background] Dale O, Nilsen T, Loftsson T, Hjorth Tonnesen H, Klepstad P, Kaasa S, Holand T, Djupesland PG. Intranasal midazolam: a comparison of two delivery devices in human volunteers. J Pharm Pharmacol. 2006 Oct;58(10):1311-8. doi: 10.1211/jpp.58.10.0003. PMID 17034653